CLINICAL TRIAL: NCT04203615
Title: Effect of Noninvasive Brain Stimulation on Hypokinetic Dysarthria and Brain Plasticity in Parkinson's Disease
Brief Title: Effect of Noninvasive Brain Stimulation on Hypokinetic Dysarthria in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masaryk University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NV16-30805A
Record Dates: First submitted 2019-12-09; First posted 2019-12-18 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: A two parallel group, randomized, placebo controlled design will be used. Twenty PD patients will be stimulated in a two weeks long therapeutical sessions (10 sessions). Other twenty PD patients will be stimulated with the same protocol using sham stimulation.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD patients with real rTMS (Active Comparator): Patients will receive real rTMS in a two weeks long sessions (10 sessions).
  Interventions: Device: Transcranial magnetic stimulation- real rTMS
- PD patients with sham rTMS (Sham Comparator): Patients will receive sham rTMS in a two weeks long sessions (10 sessions).
  Interventions: Device: Transcranial magnetic stimulation- sham rTMS

INTERVENTIONS:
Device: Transcranial magnetic stimulation- sham rTMS — Transcranial magnetic stimulation- sham figure-eight coil will be used for stimulation. This sham coil will generate only clicking noise and will not generate any magnetic field.
  Arms: PD patients with sham rTMS
Device: Transcranial magnetic stimulation- real rTMS — Transcranial magnetic stimulation- figure-eight coil will be used for stimulation. 1 Hz stimulation, 100% of Resting Motor Threshold will be used.
  Arms: PD patients with real rTMS

SUMMARY:
Hypokinetic dysarthria (HD) is common in Parkinson's disease (PD) patients and responds only partially to pharmacotherapy and surgery. The investigators will explore long-term effects of repetitive transcranial magnetic stimulation (rTMS) applied over right superior temporal gyrus, brain area known to be engaged in the feedback control of voiced speech. The project results will allow for the identification of potential therapeutic effects of rTMS as a tool that could contribute to the speech therapy of HD in PD patients. The results will also enhance our understanding of brain mechanisms underlying specific long-term effects of rTMS.

DETAILED DESCRIPTION:
A two parallel group, randomized, placebo controlled design will be used. Twenty PD patients will be stimulated in a two weeks long therapeutical sessions (10 sessions). Other twenty PD patients will be stimulated with the same protocol using sham stimulation. An MRI protocol consisting of T1, EPI BOLD, and DTI (diffusion tensor imaging) sequences and speech evaluation (acoustic signal processing and 3F test) will be performed prior to and after 10 days of rTMS and then repeated after 4, 8 and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* patients with clinically established PD (Postuma et al. 2016)

Exclusion Criteria:

* psychiatric disorders, including major depression, hallucinations
* any MRI-incompatible metal in the body
* epilepsy
* lack of cooperation
* presence of dementia

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Changes in score of the 3F Test (the unabbreviated title- "the 3F Test Dysarthric Profile") | On the beginning of the study, after completion of two weeks stimulation, 4,8 and 12 weeks after completion of stimulation sessions.
  The 3F Test Dysarthric Profile enables clinicians to characterize a wide range of signs and symptoms of dysarthria. The minimum value of this scale is 0 (anarthria), the maximum value is 90 (no disorder). Higher scores of this scale mean better outcome. This test will be administrated by speech pathologist.

SECONDARY OUTCOMES:
Resting state | On the beginning of the study, after completion of two weeks stimulation, 4,8 and 12 weeks after completion of stimulation sessions.
  The effect of stimulation on the resting state networks will be studied using fMRI measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- Central European Institute of Technology, Brno, Czechia